CLINICAL TRIAL: NCT06019026
Title: Five-year Migration Pattern and Changes in Bone Mineral Density for the Tri-Lock and Summit Femoral Stems - Radiostereometric Analysis and Dual-energy X-ray Absorptiometry of 50 Patients.
Brief Title: Five-year Migration Pattern and Bone Mineral Density for the Tri-Lock and Summit Femoral Stems.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Principal Investigator, Torben B. Hansen, Professor, MD PhD, Regional Hospital Holstebro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tri-Lock vs. Summit
Record Dates: First submitted 2023-06-13; First posted 2023-08-31 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: THA
Keywords: THA; Hip; RSA; Cementless; Radiostereometric analysis

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tri-Lock (Experimental): Total hip arthroplasty performed through posterolateral access using the uncemented Tri-Lock short stem.
  Interventions: Device: Tri-Lock
- Summit (Active Comparator): Total hip arthroplasty performed through posterolateral access using the uncemented Summit standard stem.
  Interventions: Device: Summit

INTERVENTIONS:
Device: Tri-Lock — Implant Stem
  Arms: Tri-Lock
Device: Summit — Implant Stem
  Arms: Summit

SUMMARY:
The incidence of primary hip joint prosthesis is 180 per. 100,000 inhabitants. In male patients younger than 50 years the 10-years survival of the prosthesis is 89 % and 82 % over 15 years. In women younger than 50 years the 10-years survival of the prosthesis is 87 % and 78 % over 15 years.

As revision surgery is associated with higher complication risk for the patient and poorer out-come and implant survival it is necessary to examine possible methods that may increase long-term survival of the primary hip prosthesis or facilitate better outcomes after revision of hip joint prostheses for younger patients.

In younger patients the prosthesis often is inserted without the use of cement. When not using cement, it is crucial for the final result, that there is a direct bone ingrowth of the prosthesis. The chance of getting bone ingrowth depends firstly on a good immediate mechanical fixation at surgery and secondly on osteoconductive abilities of the prosthetic surface.

This study investigates a new bone sparing implant with a new surface compared to a conventional implant.

DETAILED DESCRIPTION:
BACKGROUND

According to the Danish Hip Arthroplasty Registry 201 approximately 10.400 primary hip joint prostheses in Denmark are implanted annually, and the incidence is relatively stable. The incidence of primary hip joint prosthesis in population was 180 per. 100,000 inhabitants in 2014, with a slight predominance of female patients (60%). The average age for women is 70 and for men 67 years. Idiopathic arthritis is diagnosed in 80% of all patients receiving a hip joint prosthesis [1,2]. For older patients, the risk of later revision of a hip joint prosthesis is small. The overall survival of the primary hip joint prostheses is for all diagnoses 82% after 19 years. The prosthesis survival is poorer for younger patients, and for women. In male patients younger than 50 years the 10-years survival of the prosthesis is 89 % and 82 % over 15 years. In women younger than 50 years the 10-years survival of the prosthesis is 87 % and 78 % over 15 years. [2]. As revision surgery is associated with higher complication risk for the patient and poorer outcome and implant survival it is necessary to examine possible methods that may increase long-term survival of the primary hip prosthesis or facilitate better outcomes after revision of hip joint prostheses for younger patients.

In younger patients the prosthesis often is inserted without the use of cement. When not using cement, it is crucial for the final result, that there is a direct bone ingrowth of the prosthesis. The chance of getting bone ingrowth depends firstly on a good immediate mechanical fixation at surgery and secondly on osteoconductive abilities of the prosthetic surface. From a theoretical point of view it is also important that elastic properties of the prosthesis differ as little as possible from the elastic properties of the bone, in order to prevent a subsequent loss of bone.

INVESTIGATED IMPLANTS

The Tri-Lock femoral implant from Depuy ® is in its basic design a well-known implant that has been used since 1981 with documented good long-term results. It is an implant with bone-preserving properties and proximal coating, providing a predominantly metaphyseal anchoring. The Summit femoral implant from Depuy ®, is newer to the marked, and has a longer diaphyseal support but is predominantly metaphyseally fixed. A proximal porous implant coating will increase the surface area in contact with the metaphyseale bone and increase the coefficient of friction compared to mid-coated implants [3,4,5]. Proximal coatings may on the positive side lessen periprosthetic bone stress shielding, however, on the negative side, proximal coatings may reduce primary prosthesis fixation and lead to fibrous membrane formation with consequently implant micromotions that will eventually causing aseptic loosening of the im-plant. Hypothetical extensively coated implants have a larger porous surface and thus provide better and faster primary fixation, but there are no publications of randomized prospective clinical studies to support this. There are different porous coatings on the two investigated femoral components. Summit is coated with Porocoat porous coating, whereas Tri-Lock in the latest version is coated with the new GRIPTION technique for an even larger surface for bone ingrowth (Gription) with a new ultra-porous surface marketed as an improved immediate im-plant fixation in the bone. The total surface of the metaphyseal implant part is increased by approximately 25% with the Gription coating technique. The Gription technique may provide consistent implant seating height and additional initial stability, and these qualities may in long term ensure an improvement on implant survival.

Both femoral implants are made of Titanium. The Tri-Lock stem is designed with a reduced lateral shoulder to preserve bone in the greater trochanter, and with a shorter stem and an oblique cut stem tip, as compared to the Summit stem, in order to enhance stem insertion through minimally invasive approaches.

PRIMARY OUTCOME Mechanical loosening of a prosthesis may be suspected if the prosthesis migrates with respect to the surrounding bone [6;7]. Therefore, there is now consensus that the introduction of new implant designs including coatings and also new surgical methods should be evaluated in migration studies before they can be recommended for use in general [8;9]. Using Radiostereometric Analysis (RSA), it is now possible to get a very accurate assessment of prosthesis migration with a precision of at least 0.11 mm [10]. Clinical studies have shown that early migration of uncemented prostheses is related to the subsequent loss of the prosthesis [11;12]. For RSA tantalum beads are inserted in the prosthesis and surrounding bone. Immediately post-operatively stereoradiographs (RSA images) are made, and the initial position of the prosthesis relative to the fixed bead markers of the bone is determined. At defined time intervals new RSA images are taken. By comparison of the images the prosthesis migration in relation to the bone fixing points is determined in three dimensions, as a function of time.

Bone mineral density (BMD) around the inserted implants can be quantified by Dual Energy X-ray absorptiometry (DXA), which is an accurate method for the measurement of even small changes in BMD around femoral components [13]. DXA has been used to detect decreased bone resorption around implants with a lower stiffness [14]. A recent study from Finland demonstrated increased stem subsidence in patients with low BMD, and it is therefore advisable to screen studied patients for osteoporosis preoperatively. [15].

MATERIAL & METHODS

Design: Prospective randomized clinical study. Logistics: All newly referred patients with hip pain diagnosed with primary osteoarthritis and scheduled for hip replacement will be screened for elegibility in the study according to the study criteria. Assessed patients to be a candidate for project participation, given oral information for participants at the clinic the same day and handed over documents relating to the project. 1-2 weeks prior to surgery the patient participates in a general information session about the surgery and post-operative recovery. Here, the selected patients who wish to partici-pate in the project sign the consent form. Patients will at information day after signed consent be given an Ipad, in order to answer our questionnaires. Furthermore, there will also be conducted preoperative DXA scan.

After informed consent and using the following inclusion criteria, patients are randomized to insertion of metafysial fixed femur implant with proximal porous coating porocoat (Summit, Depuy®) or proximal Grip Tion coat (Tri-Lock, Depuy®). All patients are inserted dan same uncemented acetabular component (Pinnacle cup Depuy®). Randomization is done intraoperatively in a sealed envelope system.

RSA analysis: We will use CAD models for the femur implants, and we expect to use EGS-RSA to the acetabulum implants.

POWER:

Based on the primary endpoint (RSA) and using the following values: α= 0.05, β= 0.10 (power 90), SD = 0.6 mm, and MIREDIF: minimum relevant difference = 0.6 mm [16], sample size is 23 patients for each arm in the study.

Taking into account the risk of dropout and death in the study group inclusion is set at 25 patients per group in order to ensure that a minimum of 2 x 23 patients (46 patients) will have full follow-up of efficacy parameters at 2 years of follow-up.

ON RADIATION DOSE

Measurements were taken for the radiation dose, which shows that the stereo x-ray of the hip provides a radiation dose of 0.015 mSv [18]. This represents approximately 50% of a conventional recording of the hip. It is shown that a typical DXA measurement of the femur or spine (osteoporosis control) produce an effective dose equivalent to 0.015 mSv [19]. Conventional X-ray of the hip, gives a dose of 0.85 mSv. Normally, our hip prosthesis patients not included in this study have taken radiograph least one time within the first postoperative year. Patients in this study will have taken the same number of conventional radiographs, and in addition to 5 times DXA scan and seven times the stereoradiography. Taken from above radiation dose, patients included in this study were subjected to an additional radiation dose of 1.93 mSv. This corresponds to have taken three additional conventional radiographs of the hip, and it provides an additional risk of fatal cancer of 0.01%. This places the subjects in group IIb, where the overall risk of the irradiated individual is 1 to 10,000. [19]

REFERENCES

1. http://www.nordic.stryker.com/da/st-index-down/st_pag_patients-home/st_pag_patients-hip/st_pag_patients-hip-replacement.htm
2. Dansk Hoftealloplastik register - Årsrapport 2017
3. Cohen R. A porous tantalum trabecular metal: basic science. Am J Orthop 2002; 31(4):216-217.
4. Baad-Hansen T, Kold S, Olsen N, Christensen F, Søballe K. Excessive distal migration of fiber-mesh coat-ed femoral stems. Acta Orthop. 2011 Jun;82(3):308-14. Epub 2011 Apr 19
5. Bobyn JD, Toh KK, Hacking SA, Tanzer M, Krygier JJ. Tissue response to porous tantalum acetabular cups: a canine model. J Arthroplasty 1999; 14(3):347-354.
6. Karrholm J, Snorrason F. Subsidence, tip, and hump micromovements of noncoated ribbed femoral pros-theses. Clin Orthop 1993;(287):50-60.
7. Mjoberg B, Brismar J, Hansson LI, Pettersson H, Selvik G, Onnerfalt R. Definition of endoprosthetic loos-ening. Comparison of arthrography, scintigraphy and roentgen stereophotogrammetry in prosthetic hips. Acta Orthop Scand 1985; 56(6):469-473.
8. Malchau H. Introducing new technology: a stepwise algorithm. Spine 2000, Feb 1;25(3):285
9. Nelissen RG, Pijls BG, Kärrholm J, Malchau H, Nieuwenhuijse MJ, Valstar ER. RSA and registries: the quest for phased introduction of new implants. J Bone Joint Surg Am. 2011 Dec 21;93 Suppl 3:62-5.
10. Kiss J, Murray DW, Turner-Smith AR, Bulstrode CJ. Roentgen stereophotogrammetric analysis for as-sessing migration of total hip replacement femoral components. Proc Inst Mech Eng [H ] 1995; 209(3):169-175.
11. Karrholm J, Herberts P, Hultmark P, Malchau H, Nivbrant B, Thanner J. Radiostereometry of hip pros-theses. Review of methodology and clinical results. Clin Orthop 1997;(344):94-110.
12. Ryd L, Albrektsson BE, Carlsson L, Dansgard F, Herberts P, Lindstrand A, Regner L, Toksvig-Larsen S. Roentgen stereophotogrammetric analysis as a predictor of mechanical loosening of knee prostheses. J Bone Joint Surg Br 1995; 77(3):377-383.
13. Cohen B, Rushton N. Accuracy of DEXA measurement of bone mineral density after total hip arthro-plasty. J Bone Joint Surg Br 1995; 77(3):479-483.
14. Karrholm J, Anderber C, Snorrason F, Thanner J, Langeland N, Malchau H, Herberts P. Evaluation of a femoral stem with reduced stiffness. A randomized study with use of radiostereometry and bone densi-tometry. J Bone Joint Surg Am 2002; 84(9):1651-1658.
15. Hannu T Aro, Jessica J Alm, Niko Moritz, Tatu J Mäkinen, and Petteri Lankinen. Low BMD affects initial stability and delays stem osseointegration in cementless total hip arthroplasty in women. Acta Orthopae-dica 2012; 83 (2): 107-114
16. Onsten I, Carlsson AS, Besjakov J. Wear in uncemented porous and cemented polyethylene sockets: a randomised, radiostereometric study. J Bone Joint Surg Br 1998 Mar;80(2):345-50.
17. Valstar ER, Gill R, Flivik G, Börlin N, Kärrholm J. Guidelines for standardization of radiostereometry (RSA) of implants. Acta Orthopaedica 2006;76(4):563-572.
18. Valstar ER. Digital Roentgen Stereophotogrammetry. Development, Validation and Clinical Application. 2001.
19. Appendiks 5. Retningslinier om anvendelse af ioniserende stråling i biomedicinske forsøg. Maj 2003

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary hip osteoarthritis
2. Patients with adequate bone stock for insertion of uncemented components(no osteoporosis as assessed by pre-operative dual-energy x-ray absorptiometry (DXA) scans)
3. Informed, written consent

Exclusion Criteria:

1. Patients with neuromuscular or vascular diseases in the affected leg
2. Patients intraoperatively found unfit to uncemented components
3. Patients who can not refrain from the use of non-steroidal anti-inflammatory drugs (NSAIDs) in post-operative recovery
4. Patients with pre-operative fracture sequelae
5. Women who are, or have a wish for pregnancy during the study period.
6. Hip dysplasia or sequelae to Calves Perthes.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
Migration (3D rotation and translation) Measured with radiostereometric analysis (RSA) | 5 years
  Subsidence (distal translation mm) and retroversion (negative vertical rotation deg.)
Bone mineral density (BMD) measured with dual-energy x-ray absorptiometry | 5 years
  By Gruen zones, calculated as changes from baseline recording.

SECONDARY OUTCOMES:
Health related quality of life measured with EuroQol-5 Domain (EQ5D) | 5 years
  Patient reported outcome. Generic - calculated as normalized time trade offf score up to 1 (best)
Patient perceived hip function measured with Oxford hip score (OHS) | 5 years
  Patient reported outcome. hip-score - from 0 to 48 (best)
Pain measured on a visual analog scale (VAS) | 5 years
  active and passive measures from 0 (worst) to 10 (best)

CONTACTS AND LOCATIONS:
Overall Officials: Torben Bæk Hansen, MD, PhD, Principal Investigator — Gødstrup Hospital

IPD SHARING:
Plan to Share IPD: No
The main outcome is x-ray images and not fit for sharing due to General Data Protection Regulation (GDPR)